CLINICAL TRIAL: NCT00003704
Title: Phase I Study of Oral Capecitabine (Xeloda) as a Radiation Enhancer in Locally Unresectable, Residual, or Recurrent Colorectal Cancer Localized in the Pelvis
Brief Title: Chemotherapy Plus Radiation Therapy in Treating Patients With Unresectable, Residual, or Recurrent Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-984652; CDR0000066811 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-03-15 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
Keywords: stage III colon cancer; stage III rectal cancer; recurrent colon cancer; recurrent rectal cancer; recurrent anal cancer; stage IIIA anal cancer; stage IIIB anal cancer; stage III cervical cancer; recurrent cervical cancer; stage III ovarian epithelial cancer; recurrent ovarian epithelial cancer; stage III vulvar cancer; recurrent vulvar cancer; stage III vaginal cancer; recurrent vaginal cancer; stage III penile cancer; recurrent penile cancer; stage III endometrial carcinoma; recurrent endometrial carcinoma; stage III bladder cancer; recurrent bladder cancer; stage III malignant testicular germ cell tumor; stage III prostate cancer; recurrent prostate cancer; recurrent malignant testicular germ cell tumor; ovarian stromal cancer; recurrent urethral cancer; distal urethral cancer; proximal urethral cancer; stage III ovarian germ cell tumor; recurrent ovarian germ cell tumor; fallopian tube cancer; primary peritoneal cavity cancer; stage III uterine sarcoma; recurrent uterine sarcoma; borderline ovarian surface epithelial-stromal tumor; ovarian sarcoma
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Anus Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Ovarian Epithelial; Vulvar Neoplasms; Vaginal Neoplasms; Penile Neoplasms; Endometrial Neoplasms; Urinary Bladder Neoplasms; Testicular Neoplasms; Prostatic Neoplasms; Urethral Neoplasms; Fallopian Tube Neoplasms | interventions — Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capecitabine + radiation (Experimental): This is a dose-escalation study of capecitabine. Patients receive oral capecitabine twice a day 7 days a week for 6 weeks with concurrent radiotherapy. Radiotherapy is initiated on the same day as the initiation of capecitabine and is administered 5 days a week for 5.5-6 weeks. Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose at which 2 of 3 or 6 patients experience dose-limiting toxicity. Patients are followed every 3 months for 2 years and then every 6 months for 1 year.
  Interventions: Drug: capecitabine; Radiation: radiation therapy

INTERVENTIONS:
Drug: capecitabine
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses x-rays to damage tumor cells. Drugs such as capecitabine may make the tumor cells more sensitive to radiation therapy.

PURPOSE: Phase I trial to study the effectiveness of capecitabine in combination with radiation therapy in treating patients who have unresectable, residual, or recurrent colorectal cancer located in the pelvis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of oral capecitabine administered in combination with pelvic radiotherapy in patients with unresectable, residual, or locally recurrent cancer localized in the pelvis. II. Determine the tolerance of this regimen in these patients. III. Determine the preliminary evidence of therapeutic acticivity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of capecitabine. Patients receive oral capecitabine twice a day 7 days a week for 6 weeks with concurrent radiotherapy. Radiotherapy is initiated on the same day as the initiation of capecitabine and is administered 5 days a week for 5.5-6 weeks. Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose at which 2 of 3 or 6 patients experience dose-limiting toxicity. Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A maximum of 51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed carcinoma located in the pelvis that is unresectable, incompletely resected, or locally recurrent Must be biopsy-proven or have radiological progression All disease must be encompassable within standard pelvic radiotherapy fields No evidence of metastatic disease outside of the planned radiotherapy field

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Not specified Renal: Creatinine clearance at least 30 mL/min Other: Must maintain adequate oral nutrition (i.e., at least 1200 calories estimated intake per day) No significant infection or other concurrent medical condition that would preclude study No significant nausea or vomiting No malabsorption secondary to short-gut syndrome, Crohn's disease, or sprue No patients with more than 6 bowel movements per day or baseline no greater than grade 3 diarrhea for patients with colostomy Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for metastatic cancer At least 6 months since prior adjuvant chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior radiotherapy Surgery: At least 21 days since prior laparotomy or laparoscopic procedure with or without resection Other: No concurrent sorivudine or chemically related analogues (e.g., brivudine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 1999-04; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
overall survival | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, MD, Study Chair — Mayo Clinic
Locations (18):
- United States (17):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada